CLINICAL TRIAL: NCT02745717
Title: The Efficacy of Immunosuppressive Therapy Combined With Cord Blood Transfusion in Treatment of Severe Aplastic Anemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Ruijin Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other); Zhejiang Provincial Hospital of TCM (Other)
Responsible Party: Principal Investigator, Chun Wang, director, department of hematology, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shanghai1st-48
Record Dates: First submitted 2016-04-07; First posted 2016-04-20 (Estimated); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Severe Aplastic Anemia
Keywords: Severe aplastic anemia; immunosuppressive therapy; cord blood transfusion
MeSH Terms: conditions — Anemia, Aplastic | interventions — thymoglobulin; Antilymphocyte Serum; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cord blood and IST group (Experimental): Administration of antithymocyte ( Thymoglobulin ) 3.5mg/kg/d for 5 days, Cyclosporine Oral Product 5mg/kg/d with trough serum concentration of 200-300ng/ml, plus one unit of at least 4/6 HLA loci matched cord blood transfusion 24 hours after last dose of ATG.
  Interventions: Drug: Thymoglobulin; Procedure: Cord blood; Drug: Cyclosporine Oral Product
- IST group (Active Comparator): Antithymocyte ( Thymoglobulin ) 3.5mg/kg/d for 5 days , Cyclosporine Oral Product 5mg/kg/d with trough serum concentration of 200-300ng/ml.
  Interventions: Drug: Thymoglobulin; Drug: Cyclosporine Oral Product

INTERVENTIONS:
Drug: Thymoglobulin — administration of ATG 3.5mg/kg/d (Thymoglobuline®, Genzyme) intravenously for 5 days
  Other Names: Thymoglobuline
Procedure: Cord blood — transfusion of one unit of at least 4/6 HLA loci matched cord blood.
  Arms: cord blood and IST group
Drug: Cyclosporine Oral Product — administration of cyclosporine A 5mg/kg orally, and maintain the trough serum concentration between 200ng/ml to 300ng/ml.
  Other Names: cyclosporine A

SUMMARY:
Aim: To evaluate if additional cord blood transfusion could accelerate the hematopoietic reconstitution in severe aplastic anemia(SAA) patients receiving immunosuppressive therapy (IST).

Study design: open-labed, prospective, multicenter, randomized control study Number of subjects: 60 each group

Treatment:

IST group: ATG (Thymoglobuline®, Genzyme) 3.5mg/kg/d×5d plus oral cyclosporine A (CSA) Cord blood transfusion group: In addition to the same dose and course of ATG and CSA , one unit of cord blood having no more than 2 HLA-A, B or DRB1 mismatches is transfused 24h after last dose of ATG administration.

DETAILED DESCRIPTION:
Eligible patients should be under 60 years old with confirmed SAA, without HLA matched siblings and previous ATG treatment history. Patients will be excluded if they present any fatal disease, including respiratory failure, heart failure, liver or kidney function failure et al or severely allergic to biologic products.

To evaluate if additional cord blood transfusion could accelerate the hematopoietic reconstitution in severe aplastic anemia(SAA) patients receiving IST therapy, 120 eligible patients will be randomized to two groups, the IST group and the cord blood transfusion group. Patients in the IST group receive standard IST which including ATG (Thymoglobuline®, Genzyme) 3.5mg/kg/d×5d plus oral cyclosporine A（CSA ) started from 5mg/kg/d and adjusted to maintain trough serum concentration of 200-300ng/ml. While patients in the cord blood transfusion group receive the same dose and course of ATG and CSA as the control group and one unit of cord blood having no more than 2 HLA-A, B and DRB1 mismatches is transfused 24h after last dose of ATG administration.

The neutrophil recovery day is defined as the first day of 3 consecutive days during which the absolute neutrophil count (ANC) is >0.5×109/L, without G-CSF adminstration. Platelet recovery day is deﬁned to have occurred on the ﬁrst of 7 consecutive days with a blood platelet count (BPC) of >20×109/L, without transfusion support. Response (CR, PR or NR) is evaluated on 3, 4, 6,9, 12, 18 and 24months after treatment.

The primary end point is the neutrophil recovery day and second end points are response rate (CR+PR), treatment related mortality, disease free survival and overall survival.

.

ELIGIBILITY:
Inclusion Criteria:

1．Diagnosis of AA confirmed by bone marrow aspirate and biopsy, myelodysplastic syndrome and paroxysmal nocturnal hemoglobinuria were excluded. To confirm severe AA, the patient must fulfill at least two of the criteria: i) ANC<0.5×109/L,ii)PLT<20×109/L and iii) Ret<20×109/L ,in addition, ANC<0.5×109/L must be included.

2. Under 60 years old, male or female.

3. No HLA matched siblings.

4. No previous ATG treatment history.

5. Performance status score no more than 2 (ECOG criteria).

6．Adequate organ function as defined by the following criteria:ALT, AST and total serum bilirubin <2×ULN (upper limit of normal) Serum creatinine and BUN <1.25×ULN.

7. Adequate cardiac function without acute myocardial infarction, arrhythmia or atrioventricular block, heart failure, active rheumatic heart disease and cardiac dilatation.

8．Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment.

9. Willingness and ability to comly with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Presence of any condition inappropriate for HSCT.
2. Presence of any fatal disease, including respiratory failure, heart failure, liver or kidney function failure et al.

3．Severely allergic to biologic products.

4．Pregnancy or breastfeeding.

5．Current treatment on another clinical trail.

6．Any other condition the investigator judged the patient inappropriate for entry into this study.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
neutrophil recovery day | 5 days to 365 days
  the first day of 3 consecutive days when the absolute neutrophil count (ANC) reaches 0.5×10^9/L, without G-CSF administration .
  The day of first dose of ATG administration is record as day 0.

SECONDARY OUTCOMES:
overall response rate | 3 months to 24 months
  overall response rate is the percentage of patients who acquire complete remission and partial remission according to the criteria of British Committee for Standards in Haematology (BCSH).
overall survival | 24month
  The length of time from the start of treatment for patients with SAA are still alive.

OTHER OUTCOMES:
Treatment related mortality | 3months, 24months
  The death rate of patients because of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Chun Wang, M.D., Ph. D., Principal Investigator — Shanghai General Hospital, Shanghai Jiaotong University School of Medicine
Locations (1):
- Shanghai general hospital, Shanghai Jiaotong university school of medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Killick SB, Bown N, Cavenagh J, Dokal I, Foukaneli T, Hill A, Hillmen P, Ireland R, Kulasekararaj A, Mufti G, Snowden JA, Samarasinghe S, Wood A, Marsh JC; British Society for Standards in Haematology. Guidelines for the diagnosis and management of adult aplastic anaemia. Br J Haematol. 2016 Jan;172(2):187-207. doi: 10.1111/bjh.13853. Epub 2015 Nov 16. No abstract available. PMID 26568159
- [Background] Liu HL, Sun ZM, Geng LQ, Wang XB, Ding KY, Tang BI, Tong J, Wang ZY. Unrelated cord blood transplantation for newly diagnosed patients with severe acquired aplastic anemia using a reduced-intensity conditioning: high graft rejection, but good survival. Bone Marrow Transplant. 2012 Sep;47(9):1186-90. doi: 10.1038/bmt.2011.251. Epub 2012 Jan 16. PMID 22246086